CLINICAL TRIAL: NCT02367339
Title: Assessment of the Prevalence of Extended-Spectrum Betalactamase Producing Enterobacteriaceae Among ICU Staff
Acronym: REASSE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: University Hospital, Estaing (Other); Hopital Gabriel Montpied (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0224
Record Dates: First submitted 2015-02-12; First posted 2015-02-20 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Antibiotic Resistance; Extended-spectrum Betalactamase; Enterobacteriaceae; Escherichia Coli
Keywords: Critical Care; Nursing staff; Medical staff; Extended-spectrum betalactamase; Digestive tract colonization; Cross-contamination
MeSH Terms: conditions — Escherichia coli Infections

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Other: ESBL — Evaluation of the prevalence of ESBL-Enterobacteriaceae colonization among ICU staff

SUMMARY:
Evaluation of the prevalence of ESBL-Enterobacteriaceae colonization among ICU staff

DETAILED DESCRIPTION:
Prospective epidemiological study with voluntary non-medical staff member (i.e. nurses and nursing assistants) and medical staff in two French ICUs.

Assessment of self-reported risk factors for MDR-bacteria colonization. Self-performed rectal swab with isolation of ESBL-producting Enterobacteriaceae, identification of bacterial species and antibiotic suspectibilities.

Characterization of Escherichia coli ESBL.

ELIGIBILITY:
Inclusion Criteria:

* volunteers

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ICU staff
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Digestive tract colonization by ESBL | at day 1
  Digestive tract colonization by ESBL-producing Enterobacteriaceae on 1 faeces sample

CONTACTS AND LOCATIONS:
Overall Officials: Julien PASCAL, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France